CLINICAL TRIAL: NCT00586313
Title: Endoscopic Ultrasound(EUS)-Guided TRUCUT Biopsy (EUS-TCB) of Suspected Nonalcoholic Fatty Liver Disease(NAFLD.)
Acronym: NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0608-17
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Non-alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
Keywords: EUS Biopsy for Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- a1: Tru-Cut biopsy for liver (Experimental): Tru-Cut Biospy.
  Interventions: Device: Tru-cut biopsy; Procedure: Tru-cut

INTERVENTIONS:
Device: Tru-cut biopsy — Tru-cut biopsy may be an alternative to percutaneous and transjugular liver biopsy.
  Other Names: Wilson-Cook 19 Gauge Quick-Core EUS Biopsy Needle.
Procedure: Tru-cut — Tru-cut may be an alternative to percutaneous and transjugular liver biopsy.

SUMMARY:
Endoscopic Ultrasound involves the placement of a small flexible camera through the mouth and into the stomach to image various parts of the body. A small piece of tissue called a biopsy, of your liver nay be obtained by this method. the tissue (biopsy) would be obtained by inserting a small needle through the lining of the stomach into the liver. Consideration for this biopsy is because there may be extra fat stored within the liver. In some people who drink too much alcohol, extra fat may be stored in the liver, however, in some people who don't drink too much alcohol, this may also occur and is called :non-alcoholic fatty liver disease or NAFLD. Over time, this extra fat may lead to liver irritation and scar tissue called cirrhosis. If NAFLD is detected early enough, then treatment with medications, losing weight, or dietary changes may help avoid cirrhosis. the purpose of this study is to learn about whether doctors can obtain the biopsy from the liver by a new method. The biopsy of the liver allows the doctors to look for any signs of scar tissue or inflammation from any cause.

DETAILED DESCRIPTION:
Non-alcoholic Fatty Liver Disease (NAFLD) is an alcohol-like liver disease that occurs in individuals who do not consume excessive alcohol. Similar to alcohol-induced liver disease, NAFLD encompasses a spectrum of liver damage, ranging from non-alcoholic fatty liver (NAFL) on the most clinically benign end of the spectrum to cirrhosis on the opposite extreme where most liver-related morbidity and mortality occur. In NAFL, the liver is steatotic but generally healthy. Nonalcoholic steatohepatitis (NASH) is a more severe form of liver damage than NAFL because there is increased hepatocyte death in addition to steatosis. The liver injury in NASH triggers a repair response that sometimes leads to cirrhosis.1-3 The architecture of cirrhotic livers is distorted by regenerating nodules and fibrous tissue. Cirrhosis results when fibrosis disrupts the normal liver architecture, carving the parenchyma into nodules of hepatocytes that are separated from each other by bands of connective tissue. Some individuals with NAFLD develop cirrhosis. As in other types of liver disease, progression to this advanced stage of liver damage from NAFLD is generally thought to require many years, perhaps decades. Because most liver-related morbidity and mortality occur in cirrhotic individuals, researchers are trying to understand the basis for inter-individual differences in the tendency to develop cirrhosis. Exiting blood tests and imaging modalities have limited sensitivity for detecting liver steatosis, steatohepatitis and cirrhosis. In addition, there is no test that can distinguish NAFLD from other causes of fatty liver disease. Thus, at the present time, NAFLD is a diagnosis of exclusion.

Results from two large population-based studies are extremely useful in defining the prevalence of NAFLD in the general US adult population.4,5 The Dallas Heart Study used liver imaging to assess the prevalence of fatty liver in over 2200 adults. The overall prevalence of fatty liver in that study was 31% with a range of 24-45% of the population demonstrating hepatic steatosis. Of note, most individuals with elevated liver fat content did not demonstrate aminotransferase elevations. The latter finding helps to explain why NHANES III, another large population-based study, suggested a much lower prevalence of NAFLD in the general US adult population. In NHANES III, serum aminotransferases were used to assess NAFLD prevalence in over 15,000 adults and that approach suggested that 5.5% of the population has NAFLD. Based on the results of the Dallas Heart Study it is likely that the approach used in NHANES III underestimated the true prevalence of NAFLD in US adults. In any case, the net results from these two studies suggest that between 5.5 to 31% of the adult US population has NAFLD. To appreciate the significance of this finding, it is useful to compare the prevalence of NAFLD to that of hepatitis C, which is thought to exist in 1.8% of the US population.6 NAFLD is three to ten times more common than hepatitis C-related liver disease in the US.

Population-based studies and case series demonstrate strong associations between NAFLD and several conditions, including obesity, type 2 diabetes, and dyslipidemia, that comprise the metabolic syndrome.4,5,7-13 This suggests that the prevalence of NAFLD is likely to be much greater in these high risk populations. Studies of morbidly obese patients undergoing gastric bypass surgery support this concept. In most of these individuals, liver disease was unsuspected pre-operatively. However, intraoperative liver biopsies consistently demonstrate NAFLD. In four recent series that included over 600 subjects, the prevalence of NAFL (steatosis) ranged from 30-90% and NASH (steatohepatitis) was documented in 33-42%. Thus, over two-thirds of morbidly obese patients undergoing gastric bypass surgery have NAFL/NASH. Although overt manifestations of portal hypertension likely excluded patients as candidates for elective abdominal surgery, these four surgical series consistently identified individuals with hepatic fibrosis. Well-established cirrhosis was relatively unusual, occurring in 1-2% of the group. However, advanced fibrosis was noted in 12% and a third had unexplained periportal fibrosis. There is also a high prevalence of NAFLD is high in populations of patients with type 2 diabetes mellitus. A recent survey of 100 non-alcoholic patients with type 2 diabetes used ultrasonography to screen for NAFLD and demonstrated fatty liver in half of the group. Subsequent liver biopsy revealed NAFL in 12% and NASH in 87% of those with ultrasonographic evidence of fatty liver. Fibrosis or cirrhosis were noted in 20%.14 In patients with metabolic syndrome and hyperlipidemia, fatty liver was detected in 50% of 95 adults using ultrasonography to screen for unsuspected hepatic steatosis.15

Similar to other types of chronic liver disease, liver-related morbidity and mortality are dictated by the severity of liver damage. This concept explains observations that NAFL has a relatively benign prognosis, whereas NAFLD-related cirrhosis may be complicated by portal hypertension and hepatocellular carcinoma, eventuating in death from liver disease.2 Studies disease.2 Studies in the US and France independently demonstrated 3 easily-assessed clinical parameters that identify individuals with cryptogenic hepatitis who are likely to have advanced fibrosis on liver biopsy. These parameters are older age (greater than 45-50 years), overweight or obese body mass index, and type 2 diabetes. The probability of having bridging fibrosis or cirrhosis on liver biopsy is approximately 66% in individuals with cryptogenic hepatitis who are older and either overweight/obese or diabetic.16,17 Identification of individuals who have NASH with fibrosis has important prognostic implications. Follow-up of patients with NASH and fibrosis demonstrates that almost 30% of these individuals become cirrhotic within 5-10 years. In contrast, only about 3% of individuals with milder forms of non-alcoholic fatty liver disease develop cirrhosis after more than a decade of follow-up. Therefore, NASH with fibrosis progresses to cirrhosis both more consistently and more rapidly than simple NAFL.2,13

In order to provide optimal therapy for individuals with NAFLD, their liver disease must be diagnosed. The diagnostic evaluation of an individual who is suspected of having NAFLD has 3 goals. The first goal is to establish fatty liver disease as the etiology of the liver disease. Unfortunately, no specific serologic marker for NAFLD has been identified yet. Moreover, all of the current diagnostic tests for NAFLD have some limitation. Standard imaging tests such as ultrasonography and CT scan, may under- or over-estimate hepatic fat content.1,18 Moreover, detecting liver fat by abdominal imaging can neither distinguish alcoholic- from non-alcoholic-fatty liver disease, nor exclude other types of liver disease that might co-exist with hepatic steatosis. The second goal is to confirm the specific type of fatty liver disease, alcoholic fatty liver disease (AFLD) or non-alcoholic fatty liver disease (NAFLD). These two entities cannot be distinguished by histologic parameters but only by assessment of drinking habits of the patient. The third and arguably most important, goal of the diagnostic work-up is to establish the clinical severity and prognosis of the liver disease. Because NAFLD is common and often generates few manifestations of liver disease, it is necessary to have a high index of suspicion to identify individuals who might have NAFLD. This includes individuals with the metabolic syndrome (at least 2 of the following disorders: obesity, type 2 diabetes, hypertension and dyslipidemia) or detection of fatty liver on an imaging study of the abdomen. Imaging studies or laboratory tests may point to advanced liver disease but early cirrhosis and NAFLD without fibrosis cannot be reliably diagnosed without liver biopsy.

At this time, liver biopsy remains the "gold standard" for staging the severity of liver damage in NAFLD and all other types of chronic liver disease.2 This biopsy is traditionally performed percutaneously with or without ultrasound guidance. Needle entry for biopsy is typically into the right lobe below the diaphragm between the ribs in the right mid-axillary line. Alternatively, this may be done by an anterior approach into the left lobe. However, there are potential limitations with percutaneous biopsy including sampling error19,20 (which may not be representative of the hepatic architecture) and complications (pain, bleeding and puncture of another organ, not obtaining liver tissue). Due to anatomical considerations, some patients are not even candidates for liver biopsy by the percutaneous approach. In this case, biopsy may be performed by the transjugular method. This technique involves use of conscious sedation followed by needle access of the jugular vein. A wire is then passed through the heart and into a branch of a hepatic vein to guide a needle biopsy of the liver. Similar to percutaneous biopsy, this procedure is safe when performed by experienced operators. However, complications including neck hematoma, hepatic arteriovenous fistula, liver capsular puncture, intraperitoneal hemorrhage and death have been reported by this technique.21,22 Regardless of the approach, liver biopsy incurs monetary cost, including fees for the facility, equipment, hepatologist and pathologist, as well as for processing the tissue sample itself. On the other hand, the expense of a liver biopsy is roughly equivalent to that of magnetic resonance imaging (MRI), which is the most sensitive radiologic test for quantifying liver fat,fat; an MRI is inferior to biopsy for detecting liver inflammation and fibrosis.23

Alternative methods for acquisition of a core biopsy of the liver may be helpful in patients in whom percutaneous and transjugular liver biopsies would be difficult, risky or contraindicated. Endoscopic ultrasound (EUS)-guided fine needle aspiration (EUS-FNA) has been used for over 15 years at Indiana University Medical Center and other hospitals to sample lymph nodes and masses in the posterior mediastinum, upper abdomen and pelvis.24-29 In 2003, we published our experience of EUS-FNA of the liver using a 22-gauge needle in 77 patients without complications and to date this remains the largest series reported in the literature.30 Since that report, we have performed this procedure in over 100 patients also without a known complication (not published). In 2003, the FDA approved development of a 19-gauge Trucut biopsy (TCB) device (Wilson-Cook Medical, Inc.; Winston-Salem, North Carolina) that provides a histologic tissue sample for use with EUS. The initial reported use of this device demonstrated its safety and utility for biopsy of major upper abdominal organs (including the liver) in a swine model.31 Its subsequent use for sampling of gastrointestinal stromal tumors (GISTs), pancreatic masses and mediastinal lymph nodes in humans has also been reported.312-35 We have also studied its use in the diagnosis of nonfocal chronic pancreatitis.36 At Indiana University, we our EUS group have used this device in over 30 patients off protocol for various accepted indications without known complications (not published). The use of this EUS-TCBdevice for liver biopsy has been reported in abstract form in only two patients with suspected metastatic malignancy.37 No complications were reported in these two patients. Its use for suspected benign disease of the liver has not been reported to date.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 70 years old referred to Indiana University Hospital for outpatient upper EUS for clinical purposes (e.g., pancreatic disease).
2. Increased hepatic enzymes (AST or ALT) above the upper limit of normal within the past 3 months. These values at University Hospital are ALT>45 U/L and AST> 41 U/L but may vary among laboratories at different institutions.
3. Evidence of fatty liver (as detected by an increase in echogenicity or brightness of the liver) by EUS exam.
4. Liver biopsy for suspected NAFLD is clinically indicated as determined by Dr Naga Chalasani, one of our staff hepatologists who is an expert in NAFLD.

Exclusion Criteria:

1. Inpatient status.
2. Normal liver enzyme tests (AST, ALT).
3. Previous or current alcohol abuse (≥3 drinks/day for men; ≥2 drinks/day for women)
4. Planned liver biopsy within 30 days for known or suspected liver disease.
5. Suspected metastatic lesion in the liver by any previous imaging study or discovered during EUS exam.
6. EUS-FNA of the liver is required for another reason (i.e. suspected metastatic lesion)
7. Newly diagnosed, currently treated or suspected malignancy. (In this case, the diagnosis of NAFLD would not likely impact patient care or survival). Patients with a previously diagnosed malignancy that is in remission will be considered eligible.
8. Previously diagnosed NAFLD including steatosis or NASH (in this situation, another biopsy is not beneficial to the patient).
9. Chronic liver disease including Hepatitis B, Hepatitis C, Wilson's disease, alpha-1-antitrypsin disease, autoimmune hepatitis.
10. Known or suspected cirrhosis.
11. Esophageal or gastric varices by previous imaging or discovered during EUS.
12. Previous liver surgery including resection or transplant.
13. Thrombocytopenia (platelets <150,000)
14. Anemia (hemoglobin <10 gm/dL).
15. Coagulopathy (INR>1.2 or aPTT > 35 secs).
16. Use of coumadin or other anticoagulants.
17. Use of aspirin or nonsteroidal antinflammatory product within 7 days of EUS.
18. Total bilirubin >2.0 mg/dL and dilated bile duct on previous imaging study.
19. Inability to provide informed consent.
20. Pregnancy or suspected pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. DeWitt, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dewitt J, McGreevy K, Cummings O, Sherman S, Leblanc JK, McHenry L, Al-Haddad M, Chalasani N. Initial experience with EUS-guided Tru-cut biopsy of benign liver disease. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):535-42. doi: 10.1016/j.gie.2008.09.056. PMID 19231495
- [Derived] Sey MS, Al-Haddad M, Imperiale TF, McGreevy K, Lin J, DeWitt JM. EUS-guided liver biopsy for parenchymal disease: a comparison of diagnostic yield between two core biopsy needles. Gastrointest Endosc. 2016 Feb;83(2):347-52. doi: 10.1016/j.gie.2015.08.012. Epub 2015 Aug 13. PMID 26278654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive subjects undergoing EUS with suspected hepatic parenchymal disease
Groups:
- EUS Tru-cut Biopsy: Transgastric EUS-TCB may prove to be a safe alternative to percutaneous and transjugular liver biopsy methods in obtaining liver biopsy samples.
  EUS Tru-cut biopsy: Transgastric EUS-TCB may prove to be a safe alternative to percutaneous and transjugular liver biopsy methods in obtaining liver biopsy samples. This technique may be particularly helpful to obtain liver biopsies in patients with morbid obesity or patients in whom there is no obtainable view to obtain a percutaneous biopsy.
Period: Overall Study
Arm/Group | EUS Tru-cut Biopsy
Started | 21
Completed | 19
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: 13 females
Groups:
- Participants Undergoing the Tru-Cut Biopsy: Transgastric EUS-TCB may prove to be a safe alternative to percutaneous and transjugular liver biopsy methods in obtaining liver biopsy samples.
  EUS Tru-cut biopsy: Transgastric EUS-TCB may prove to be a safe alternative to percutaneous and transjugular liver biopsy methods in obtaining liver biopsy samples. This technique may be particularly helpful to obtain liver biopsies in patients with morbid obesity or patients in whom there is no obtainable view to obtain a percutaneous biopsy.
Arm/Group | Participants Undergoing the Tru-Cut Biopsy
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Median Total Specimen Length
Description: Median Total Specimen Length grouped for indication for liver biopsy: Suspected NAFLD, Intrahepatic Cholestasis, Exclusion of Cirrhosis, Increased Liver Function Tests (LFTs) of Uncertain Cause and the Total.
Time Frame: 24 months
Measure: Median (Full Range); unit: mm
Arm/Group | EUS Tru-cut Biopsy
Number analyzed (Participants) | 21
mm
  Suspected NAFLD, n=9 | 8 [1 to 13]
  Intrahepatic Cholestasis, n=4 | 14 [3 to 22]
  Exclusion of Cirrhosis, n=4 | 8 [6 to 22]
  Increased Liver Function Tests (LFTs), n=4 | 11.5 [6 to 23]
  Total, n=21 | 9 [1 to 23]

2. Secondary Outcome: The Number of Procedural Complications
Description: Major procedural complications could include: hospitalization, surgery or a radiologic procedure to correct an adverse event; bleeding, infection. Minor procedural complications could be increase in abdominal pain, self-limited hypoxia, bradycardia, tachycardia, hypo or hyper-tension, change in vital signs.
Time Frame: 24 months
Measure: Number; unit: complications
Arm/Group | EUS Tru-cut Biopsy
Number analyzed (Participants) | 21
complications | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | EUS Tru-cut Biopsy
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
The small sample size and low-risk population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes